CLINICAL TRIAL: NCT02844309
Title: The Efficacy of Thalidomide Plus Cyclophosphamide and Dexamethasone Following by Thalidomide and Prednisone Maintenance Therapy for the Newly Diagnosed Waldenström Macroglobulinemia - a Prospective Multicentre Phase Ⅳ Trial From China
Brief Title: The Efficacy of TCD Following by TP Maintenance Therapy in Newly Diagnosed WM
Acronym: BDH-WM02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015004
Record Dates: First submitted 2016-07-17; First posted 2016-07-26 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Waldenström Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide (Experimental): thalidomide 50-150mg per night
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — thalidomide 50-150 mg per night
  Other Names: Thal

SUMMARY:
The purpose of this study is to evaluate the efficiency of an oral regimen in newly diagnosed Waldenström macroglobulinemia: thalidomide plus cyclophosphamide and dexamethasone following by thalidomide and prednisone maintenance therapy.

DETAILED DESCRIPTION:
Enrolled patients will accept maximum 8 cycles of thalidomide plus cyclophosphamide and dexamethasone. if a partial remission response or better is achieved, thalidomide plus prednisone maintenance therapy will be given for no more than two years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >=18 years
2. diagnosed with WM
3. Untreated or mild treated without standard regimens,especially untreated with rituximab and/or bortezomib
4. symptom patients
5. with life-expectancy more than 3 months.

Exclusion Criteria:

1. diagnosed with other malignancies outside B-NHL within one year(including active centre neural system lymphoma)
2. Transformed lymphoma
3. liver or renal function lesion unrelated to lymphoma
4. serious complications such as uncontrolled diabetes,gastric ulcer or other serious angiocardiopathy determined by the physician
5. HIV positive or active HBV infection or other uncontrolled systematic infection
6. clinical central nervous dysfunction
7. serious surgery within 30 days
8. pregnancy or baby nursing period or un-contracepted child-bearing period woman;
9. allergy to the trail drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 12 months

SECONDARY OUTCOMES:
progress-free survival | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Doc, Principal Investigator — institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Shuhua Yi, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided
whether to publish primary data is dependent on the local law